CLINICAL TRIAL: NCT05995860
Title: Pilot Study of a Rapid Triadic Communication Intention Elicitation Intervention (PRECursOr) to Improve Supportive Oncology Care Delivery for Patients With Advanced, Incurable Cancer and Their Caregivers
Brief Title: Study of a Rapid Triadic Communication Intention Elicitation Intervention to Improve Supportive Oncology Care Delivery
Acronym: PRECursOr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kristin Levoy, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO-IUSCCC-0827
Record Dates: First submitted 2023-07-10; First posted 2023-08-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Vulvar Cancer; Ovarian Cancer; Uterine Cancer; Vaginal Cancer
MeSH Terms: conditions — Vulvar Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Vaginal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group triads (No Intervention)
- Intervention group triads (Experimental)
  Interventions: Behavioral: Intervention group triads

INTERVENTIONS:
Behavioral: Intervention group triads — The intervention consists of a rapid (less than 10-minute) communication intention elicitation exercise (via Freelisting), which is conducted independently with the patient, caregiver, and provider immediately prior to the outpatient oncology encounter. Patients, caregivers, and providers will not be instructed to endorse the Freelist responses that were generated by the intervention prior to the outpatient encounter-leaving the decision to discuss elicited communication intentions during the encounter up to individuals as the conversation naturally occurs. As with the control group, post-encounter survey data will also be collected independently from the patient, caregiver, and the provider, followed by a post-encounter qualitative interview conducted jointly with the patient and caregiver.
  Other Names: PRECursOr
  Arms: Intervention group triads

SUMMARY:
The purpose of this study is to help test an idea designed to foster more supportive talk between providers (doctors or nurse practitioners), patients, and caregivers during an outpatient oncology appointment. A caregiver is the person the patient identifies is primarily involved in their healthcare. This study is collecting your reaction to this idea in order to understand needed changes before we introduce the idea to a larger group of patients.

DETAILED DESCRIPTION:
This pilot study focuses on an intervention (freelisting) designed to elicit supportive oncology communication intentions among the patient-caregiver-provider triad prior to an outpatient oncology encounter. The goal is to shape communication behaviors during the encounter to improve outcomes of the encounter.

ELIGIBILITY:
Inclusion Criteria:

* patients will:

  1. be adult women with an incurable gynecologic cancer (i.e., evidence of refractory/progressive disease after first-line treatment or recurrent disease),
  2. not be receiving specialty palliative care or hospice,
  3. read/speak English, and
  4. be able to provide written informed consent.
* caregivers will:

  1. identify as the individual who is primarily involved in the patient's care,
  2. be able to attend the oncology encounter,
  3. read/speak English, and
  4. be able to provide written informed consent.
* providers will:

  1. specialize in gynecologic oncology, and
  2. provide outpatient care at IUSCCC gynecologic oncology clinic.

Exclusion Criteria:

patients and/or caregivers will be excluded if either one or both demonstrate:

1. cognitive impairment, or
2. speech/hearing difficulties precluding participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Evaluate overall recruitment rates. | Once all surveys in the sample size are completed, 9 months anticipated
  PRECursOr will meet or exceed feasibility (overall recruitment, recruitment rate, measure completion, encounter duration).
Evaluate overall participant satisfaction surveys. | Once all surveys in the sample size are completed, 9 months anticipated
  PRECursOr will meet or exceed acceptability (satisfaction, acceptability of approach) benchmarks per patient and caregiver questionnaire.
Explore group differences in communication behaviors during the audio-recorded encounters. | Once all encounters in the sample size are completed and transcribed, 9 months anticipated
  The intervention group will demonstrate increased communication behaviors during the encounter (i.e., breadth of supportive oncology domains discussed) and a trend toward greater benefits in the immediate (e.g., quality of communication) and proximal (e.g., shared understanding of treatment goals, distress, anxiety) outcomes of communication.
Explore group differences in exit interview outcomes following the encounters. | Once all encounters in the sample size are completed and transcribed and survey/interview completion, 9 months anticipated
  The intervention group will demonstrate increased communication behaviors and a trend toward greater benefits in the immediate (e.g., quality of communication) and proximal (e.g., shared understanding of treatment goals, distress, anxiety) outcomes of communication.
Identify intervention approaches in exit interview that contributed to positive and/or negative outcomes | Once all surveys in the sample size are completed, 9 months anticipated
  Identify intervention approaches that contributed to positive and/or negative outcomes to inform intervention refinement using qualitative research methods.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No